CLINICAL TRIAL: NCT02989519
Title: Comparison of the Efficacy of Oral Progesterone and Vaginal Progesterone After Tocolytic Therapy in Threatened Preterm Labor
Brief Title: Efficacy of Oral Progesterone and Vaginal Progesterone After Tocolytic Therapy in Threatened Preterm Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanpasitthiprasong Hospital (Other Government)
Responsible Party: Principal Investigator, Piyawadee Wuttikonsammakit, Instructor, Sanpasitthiprasong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SPS2016-01
Record Dates: First submitted 2016-12-07; First posted 2016-12-12 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Preterm Delivery
Keywords: preterm labor; progesterone efficacy; threatened preterm labor
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Dydrogesterone; Progesterone; Utrogestan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no progesterone (No Intervention): All women with preterm labor underwent standard tocolysis, which was administered for at least 48 hours, to allow corticosteroid promote fetal lung maturation
- oral progesterone (Experimental): All women with preterm labor underwent standard tocolysis, which was administered for at least 48 hours, to allow corticosteroid promote fetal lung maturation. All women in this arm received oral progesterone (dydrogesterone 10 mg; Duphaston™) per oral three times a day
  Interventions: Drug: dydrogesterone
- vaginal progesterone (Experimental): All women with preterm labor underwent standard tocolysis, which was administered for at least 48 hours, to allow corticosteroid promote fetal lung maturation. All women in this arm received vaginal progesterone (micronized progesterone 200 mg; Utrogestan™) at bed time.
  Interventions: Drug: Micronized progesterone

INTERVENTIONS:
Drug: dydrogesterone
  Other Names: Duphaston
  Arms: oral progesterone
Drug: Micronized progesterone
  Other Names: Utrogestan
  Arms: vaginal progesterone

SUMMARY:
The purpose of this study is to determine efficacy of vaginal and oral progesterone after tocolytic therapy in threatened preterm labor

DETAILED DESCRIPTION:
A randomized controlled trial was conducted from August 2015 through December 2016. All pregnant women with single pregnancies of 28 to 33 weeks and 6 days who had been experienced for threatened or preterm labor with intact membrane as in inclusion criteria were approached and ask for enrollment. The gestational age of all patients was confirmed by antenatal record review and ultrasonographic confirmation. Threatened preterm labor was defined as the presence of regular uterine contractions without significant cervical changes as determined by digital pelvic examination. Preterm labor was defined as the simultaneous presence of regular uterine contractions and cervical changes, shortening and/or softening, or dilatation, as determined by digital pelvic examination. The women with preterm labor underwent standard tocolysis, which was administered for at least 48 hours, to allow corticosteroid promote fetal lung maturation. The patients who had proven membranes ruptured, and ultrasonographically found placenta previa, multiple pregnancy, fetal anomaly or aneuploidy would excluded. The participants had emergency condition that required for emergency delivery such as fetal distress, chorioamnionitis were also excluded. Participants were randomized into three groups which generated by computer programme to receive whether oral progesterone (dydrogesterone 10 mg; Duphaston™) per oral three times a day or vaginal progesterone (micronized progesterone 200 mg; Utrogestan™) or no progesterone (controlled group). All patients were digitally pelvic examined for evaluation of Bishop score and assessed cervical length by transvaginal ultrasound at enrollment and follow up visit at two weeks apart. Cervical length was measured by standard technique with a covered probe inserted into vagina after each woman had emptied her bladder. Excessive pressure on cervix was avoided. The mean value of 3 consecutive measurements was used for analysis. Informed consent and demographic data were obtained at the enrollment. Primary outcomes were preterm delivery before 34 and 37 weeks. Secondary outcomes include time until delivery (latency period,days), change of cervical length (cervical attenuation), maternal outcome, neonatal outcome, and side effects of drugs were collected. The main outcomes of preterm delivery, gestational age at parturition and birthweight were also collected by telephone call in case of out-side-hospital born or in case loss to follow up. Monitoring of all patients was evaluated every follow up visit for drug side effect, allergic response, and adverse events Statistical analysis Sample size was calculated according to the results of two studies by Dorota AgataBomba - Opon and Manju Choudhary which showed significant decreased preterm delivery <34 weeks (9.8% vs 35.3%,p=0.002) in vaginal progesterone group, and significant decreased preterm birth (33% vs 58% ; p= 0.034) in oral progesterone group. The sample size of 231 was used to evaluate the primary outcome of both drugs. Descriptive statistics were carried out using mean, median, standard deviation, interquartile range. Categorical data were tested for significance with the χ2tests. Continuous data were evaluated for normal distribution and tested for significance with ANOVA and Kruskal-Wallis test. Student t test and Man-Whitney U test were used to test significance between groups in case there is significant detection in ANOVA and Kruskal-Wallis test among groups. Statistical significance was defined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancies of 28 to 33 weeks and 6 days who had been experienced for threatened or preterm labor with intact membrane

Exclusion Criteria:

* Proven membranes ruptured
* Ultrasonographically found placenta previa, multiple pregnancy, fetal anomaly
* Aneuploidy detected.
* Had emergency condition that required for emergency delivery such as fetal distress, chorioamnionitis, prolapsed cord

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
preterm delivery before 34 and 37 weeks | 3 months

SECONDARY OUTCOMES:
change of cervical length | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Piyawadee Wuttikonsammakit, MD, Principal Investigator — Instructor
Locations (1):
- Piyawadee Wuttikonsammakit, Nai Muang, Changwat Ubon Ratchathani, Thailand

IPD SHARING:
Plan to Share IPD: No